CLINICAL TRIAL: NCT05968339
Title: Survey Evaluating Elements in Choosing Mentors/ Mentees in Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: AZ Sint-Lucas Brugge (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Staff, Université Libre de Bruxelles
Other Study IDs: Mentor-Anesth
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — The survey will be distributed via scientific anesthesiology societies and will be open for a total of 12 consecutive months.
  Participation in the survey will be voluntary and anonymous - individual consent will be implied by willingness to complete the survey.
  The survey will be conducted via SurveyMonkey. SurveyMonkey allows "Health Insurance Portability and Accountability Act" (HIPAA)(12) compliant surveys to be created. These follow strict rules around the protection of health information. Of note, SurveyMonkey is also GDPR (General Data Protection Regulation) compliant.
  Data gathered from the questionnaires will be safely stored. Access to the database will be password protected and only the authors will have access for the purpose of data analysis at the end of the survey period. Analysis using chi squared tests and logistic regressions will be performed by trained statisticians.

SUMMARY:
Mentorship is increasingly recognised as a core component of career advancement, medical education and psychosocial support.

Mentorship is defined as the relationship between a mentor and a mentee, where both collegially gain from an open and active relationship

Overall, there is little known about mentorship in anaesthesia.

To our knowledge, no study has yet explored the fostering of an anaesthetic mentor-mentee relationship from the point of view of the mentor and mentee themselves. Preferences with regards to implementation programs versus free choice and the importance of sociodemographic characteristics (gender, ethnicity, sexuality, disability, age) have also yet to be investigated.

The prevalence of mentor-mentee relationships/ the understanding of mentor and mentee choice in anaesthesia will be studied.

In parallel, key socio-demographics that are linked to the choice of mentor-mentee, as well as evaluate availability of mentors, and other barriers to finding mentorship will also be investigated.

Hypothesis: mentorship might be affected by demographics such as gender, age, ethnicity, working country, experience, academia and subspecialty.

DETAILED DESCRIPTION:
Mentorship is increasingly recognised as a core component of career advancement, medical education and psychosocial support.

Mentorship is defined as the relationship between a mentor and a mentee, where both collegially gain from an open and active relationship.

A mentor can be seen as a role model, a supervisor, an advisor, and a career coach.

A mentee is counselled, trained, or advised by a mentor and can be assimilated to a protégé.

A mentee has the potential to gain multiple advantages from their mentorship such as protection, sponsorship, exposure, promotion and transmission of professional ethics.

Moreover, psychosocial support in the form of identity fostering, sense of competence and role effectiveness might protect the mentee from burdens such as burnout. As a mentee's needs often change over the course of their career, it is therefore possible to have multiple mentors at different stages.

When engaging in an mentoring relationship, free choice has been shown to be more effective than automatic assignment. Unfortunately, free choice can enhance inequities in mentorship as various groups lack representation, social connections and experience a lack of opportunities to find the right mentor. Gender inequities in finding mentorship have been reported and may affect job satisfaction and career advancement.

When establishing mentorship, it is important to foster trust. Even though free choice has been reported as essential, some mentoring programs (endorsed by societies such as ESAIC / ASA) have been successfully implemented within anaesthesia(6). Sub-societies, such as ASRA, have established well-defined mentor/mentee programs (ASRA Pain Medicine Mentor Match program) where mentor/ mentee match is based on common interests.

However, there is overall little known about mentorship in anaesthesia.

A survey of mentorship in Canadian anaesthesiology residents reported multiple barriers to successful mentorship: time constraint, personal or professional incompatibility (in mentorship programs) and lack of resident choice in mentor selection(3).

A qualitative study of perceptions of mentorship by both faculty and residents identified the following:

* Evolution of the mentor-mentee relationship during residency from a primary focus on psychosocial aspect to a need of career facilitation in the end.
* Importance of congruence/ representation of gender, culture and ethnicity.

An anaesthesia specific survey has already investigated the practices of mentorship and career development during residency in the USA from the point of view of program directors.

To our knowledge, no study has yet explored the fostering of an anaesthetic mentor-mentee relationship from the point of view of the mentor and mentee themselves. Preferences with regards to implementation programs versus free choice and the importance of sociodemographic characteristics (gender, ethnicity, sexuality, disability, age) have also yet to be investigated.

The prevalence of mentor-mentee relationships/ the understanding of mentor and mentee choice in anaesthesia will be studied.

In parallel, key socio-demographics that are linked to the choice of mentor-mentee, as well as evaluate availability of mentors, and other barriers to finding mentorship will also be investigated.

Hypothesis: mentorship might be affected by demographics such as gender, age, ethnicity, working country, experience, academia and subspecialty.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists who are members of ESAIC/ASA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey will be distributed via anesthesiology societies (ESAIC: European Society of Anaesthesiology and Critical Care and ASA: American Society of Anesthesiologists).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Survey-1 | 12 months
  The first part of the survey consists of sociodemographic data.
Survey-2 | 12 months
  The second part evaluates preferences choosing a mentor/ a mentee, as well as facilitators and barriers to mentorship relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Saxena, MD; PHD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- AZ Sint Jan Brugge, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gisselbaek M, Marsh B, Soriano L, Jackman S, Seidel L, Albert A, Matot I, Coppens S, Narouze S, Barreto Chang OL, Saxena S. Gender and Race/Ethnicity dynamics in anesthesiology mentorship: results of a European survey. BMC Anesthesiol. 2024 Sep 6;24(1):311. doi: 10.1186/s12871-024-02692-6. PMID 39242999